CLINICAL TRIAL: NCT04908579
Title: Efficacy of Preventive Ketamine on Postoperative Pain: A Randomized, Double-blind Trial of Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Efficacy of Preventive Ketamine on Postoperative Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD 87/ 2021
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- - GROUP (I): 30 patients (Active Comparator)
  Interventions: Drug: bupivacaine(intraperitoneally) and ketamine (intraperitoneally)
- - GROUP (II): 30 patients (Active Comparator)
  Interventions: Drug: bupivacaine(intraperitoneally) and ketamine (intravenously)
- - GROUP (III) (Control): 30 patients (Active Comparator)
  Interventions: Drug: bupivacaine(intraperitoneally)

INTERVENTIONS:
Drug: bupivacaine(intraperitoneally) and ketamine (intraperitoneally) — 1. 40 ml volume of bupivacaine 0.25% + ketamine 0.5 mg/kg distributed as 30 ml intraperitoneally and 10 ml as port site infiltration
  2. 10 ml normal saline 0.9% will be given intravenous.
  Arms: - GROUP (I): 30 patients
Drug: bupivacaine(intraperitoneally) and ketamine (intravenously) — 1. 40 ml volume of bupivacaine 0.25% only distributed as 30 ml intraperitoneally and 10 ml as port site infiltration
  2. 10 ml volume of ketamine 0.5 mg/kg intravenously will be given after delivering the gastric sleeve and before start closure of port sites.
  Arms: - GROUP (II): 30 patients
Drug: bupivacaine(intraperitoneally) — 1. 40 ml volume of bupivacaine 0.25% only distributed as 30 ml intraperitoneally and 10 ml as port site infiltration
  2. 10 ml normal saline 0.9% will be given intravenous.
  Arms: - GROUP (III) (Control): 30 patients

SUMMARY:
* Although bariatric surgery is mainly performed laparoscopically, analgesic optimization is still essential to reduce complications and to improve the patients' comfort. In laparoscopic sleeve gastrectomy, the intraoperative peritoneal instillation of bupivacaine hydrochloride (30 ml, 0.25%) was known to be safe and effective in reducing postoperative pain, nausea, and vomiting.
* Furthermore, usage of ketamine both as a pre and post-operative pain management is well established. Ketamine can be used solely or in combination with other co-adjuvant drugs, increasing their efficacy. Many therapeutic properties of ketamine have been attributed to its antagonism mechanism to N-Methyl-D-aspartate receptors.

ELIGIBILITY:
Inclusion Criteria:

* - Body mass index > 35 and < 60 kg/m2
* Either medically free or with well controlled hypertension and/or diabetes.

Exclusion Criteria:

* - Patient's refusal to participate in the study
* BMI > 60 kg/m2.
* Age less than 21 years.
* Patients with severe systemic disease which is not life-threatening.
* Patients on antipsychotics, antidepressants and/or corticosteroids.
* Patients with history of obstructive sleep apnea.
* Allergic reaction to any of the study medications.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to first given rescue analgesia(minutes) | 24 hours postoperatively
  Time to first given rescue analgesia(minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No